CLINICAL TRIAL: NCT00552084
Title: Fish Oil for Atrial Fibrillation - Effect and Mechanisms
Brief Title: Evaluating the Effectiveness of Fish Oil Supplements at Reducing the Recurrence of Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); eCardio Diagnostics (Unknown); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine, Professor of Pharmacology, Assistant Director of the Division of Clinical Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 543; R01HL087254 (NIH); HL 087254
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Atrial Fibrillation
Keywords: Fish Oil
MeSH Terms: conditions — Atrial Fibrillation | interventions — Fish Oils; Omacor; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish Oil (Experimental): 4 grams fish oil daily for 24 weeks
  Interventions: Drug: Fish oil
- Placebo (Placebo Comparator): corn oil taken daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fish oil — Fish oil supplements 4 gms will be taken daily for 24 weeks.
  Other Names: Lovaza capsule (1 gm)containing 465 mg EPA and 375 mg DHA.
  Arms: Fish Oil
Drug: Placebo — Placebo supplements will be taken daily for 24 weeks.
  Other Names: Corn oil
  Arms: Placebo

SUMMARY:
Atrial fibrillation (AF) is a heart rhythm disorder that usually involves a rapid heart rate. People who take fish oil supplements may reduce the risk of a recurrence of AF. This study will evaluate the effectiveness of fish oil at decreasing the recurrence of AF and will examine the reasons why fish oil may reduce this risk.

DETAILED DESCRIPTION:
AF is the most common type of serious heart arrhythmia. It affects approximately 2% of the population and is becoming more common. In AF, the heart's atria, or upper chambers, contract in a very disorganized and abnormal manner and are unable to correctly pump blood into the heart's ventricles, or lower chambers. Symptoms may include a rapid or irregular pulse, dizziness, fainting, or breathing difficulty. Recent studies suggest that inflammation plays a fundamental role in the development of AF. Inflammation, and the resulting oxidative stress, can cause cellular and tissue damage. In turn, this may alter heart function, potentially leading to both the onset and recurrence of AF. Markers of inflammation, such as C-reactive protein (CRP) and interleukin-6 (IL-6), are often elevated in patients with AF, providing further evidence of inflammation's role. While there are several treatment options for AF, they are usually only moderately effective. Previous research has shown that fish oil supplements have anti-inflammatory, antifibrotic, and antioxidant effects and can reduce the risk of AF following surgery. However, it is not known exactly how fish oil reduces this risk and whether the same positive effect will carry over in people who experience the more common type of AF that is unrelated to surgery. The purpose of this study is to evaluate the effectiveness of fish oil supplementation at decreasing the recurrence of AF in adults who have not undergone recent surgery. Researchers will also examine the ways in which fish oil reduces AF recurrence.

This study will enroll people who have had at least two occurrences of AF. Participants will be randomly assigned to receive either fish oil supplements or placebo for 24 weeks. At study visits at baseline and Weeks 2, 4, 8, 12, 18, and 24, participants will undergo a medical and social history review, a physical exam, and blood and urine collection. At the baseline study visit, an electrocardiogram will also occur.

ELIGIBILITY:
Inclusion Criteria:

* >=21 years of age
* a history of atrial fibrillation
* a history of at least two occurrences of atrial fibrillation or atrial flutter, at least one of which is atrial fibrillation
* an electrocardiogram that was recorded within 12 months of randomization showing atrial fibrillation or atrial flutter
* sinus rhythm at the time the first dose of randomized medication is taken
* stable antiarrhythmic medications
* if the patient has had an ablation for atrial fibrillation or flutter or a MAZE procedure, the qualifying episode of atrial fibrillation must have occurred at least 3 months post-procedure
* normal serum potassium level within the last 28 days
* provided informed consent

Exclusion Criteria:

* permanent atrial fibrillation or flutter
* New York Heart Association class III or IV heart failure or Canadian Cardiovascular Society class III or IV angina pectoris
* cardiac or thoracic surgery within the previous 3 months
* acute pericarditis within the previous 3 months
* other reversible causes of atrial fibrillation such as thyrotoxicosis
* acute myocardial infarction or unstable angina within the previous 3 months
* history of neurologic event (TIA or stroke)within the past 3 months
* history of acute congestive heart failure precipitated by atrial fibrillation, and the patient is not receiving rate-control therapy
* Wolff-Parkinson-White syndrome
* a medical condition that is likely to be fatal in less than one year
* active, uncontrolled co-morbid inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease, SLE)
* receiving cytotoxic chemotherapy or radiotherapy for cancer
* taking a fish oil supplement
* allergic to fish
* bleeding event not related to trauma or surgery requiring hospitalization or transfusion in previous year
* systolic blood pressure < 90 mm Hg or heart rate <50 beats/minute
* history of ventricular fibrillation or sustained ventricular tachycardia, or presence of an implanted defibrillator placed for the occurrence of such an event or the presence of an Implantable Cardioverter-Defibrillator (ICD) that has discharged appropriately for a ventricular arrhythmia
* pregnant or breast feeding
* enrollment in another research study involving an intervention
* on dialysis or recipient of a renal transplant
* use of potentially cardiotoxic illegal drugs (cocaine, methamphetamine, opioids) in the last 12 months
* Treated for alcoholism and currently drinking alcohol to excess or alcoholic cardiomyopathy as the primary clinical diagnosis and currently drinking alcohol to excess
* presence of an iron-storage disease, such as hemochromatosis, transfusional hemosiderosis, or those subjects in whom a daily dose of up to 20 mg elemental iron (in and of itself or in addition of current iron supplementation) would post a risk for toxicity from iron overload
* subjects receiving or anticipated to receive intravenous iron therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2007-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Stein, Principal Investigator — Vanderbilt Medical School
Locations (1):
- Vanderbilt Medical School, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Vanderbilt C, Free M, Li J, Gebretsadik T, Bian A, Shintani A, McBride BF, Solus J, Milne G, Crossley GH, Thompson D, Vidaillet H, Okafor H, Darbar D, Murray KT, Stein CM. Effect of omega-three polyunsaturated fatty acids on inflammation, oxidative stress, and recurrence of atrial fibrillation. Am J Cardiol. 2015 Jan 15;115(2):196-201. doi: 10.1016/j.amjcard.2014.10.022. Epub 2014 Oct 29. PMID 25465932

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 4 medical centers in Nashville Tennessee, and at the Marsh field Clinic in Madison, Wisconsin. Between December 2007 and December 2012, 241 patients were enrolled and 190 (178 at Vanderbilt, 12 at other sites) were randomized to fish oil (126) or placebo (64). Of 190 enrolled, 173 (91%) completed the study.
Pre-assignment Details: Patients were >= 21 years old with a history of at least 2 occurrences of atrial fibrillation or atrial flutter, and in sinus rhythm at randomization. Randomization was performed according to a computer-generated block scheme according to anti-arrhythmic therapy: 1. no therapy, 2. amiodarone, 3. class 1 anti-arrhythmic drugs, 4.sotalol/dofetilide.
Period: Overall Study
Arm/Group | Fish Oil | Placebo
Started | 126 | 64
Completed | 118 | 55
Not Completed | 8 | 9
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — change in anti-arrythmic drug | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil | Placebo | Total
Number analyzed (Participants) | 126 | 64 | 190
Age, Continuous [Mean (Full Range); unit: years] | 61.9 [21 to 82] | 61.5 [28 to 82] | 61.7 [21 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 38 | 100
  >=65 years | 64 | 26 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 22 | 81
  Male | 67 | 42 | 109
Region of Enrollment [Number; unit: participants]
  United States | 126 | 64 | 190

OUTCOME MEASURES:

1. Primary Outcome: Documented Recurrence of Atrial Fibrillation/Atrial Flutter
Description: Trans-telephonic electrocardiographic monitoring (TTM) device were used to send transmissions every 2 weeks and each time a participant had symptoms suggestive of arrhythmia.
Time Frame: Measured at Week 24 or exit
Measure: Number; unit: percentage of participants
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 126 | 64
percentage of participants | 59 | 47

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 24 week study, after participants took first dose of study medication or placebo.
Arm/Group | Fish Oil | Placebo
Serious Adverse Events (participants affected / at risk) | 2/126 | 3/64
Other Adverse Events (participants affected / at risk) | 40/126 | 13/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil (N=126) | Placebo (N=64)
pseudogout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
rapid atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fish Oil (N=126) | Placebo (N=64)
Low INR (Blood and lymphatic system disorders) | 17 | 2
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Diarrhea (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 6 | 2

LIMITATIONS AND CAVEATS:
We determined recurrence of Atrial Fibrillation(AF) by both routine and symptomatic TTM transmissions. We did not examine the effect of therapy on total AF burden. Sample size was relatively small, and included a heterogeneous patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes